CLINICAL TRIAL: NCT00586742
Title: SLAP Lesions; a Comparison of Conservative and Operative Treatment. A Prospective, Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00001870
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: SLAP Lesions
Keywords: SLAP lesions; labral repair; bicepstenodesis; conservative treatment
MeSH Terms: interventions — Suture Anchors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Labral repair with suture anchors
  Interventions: Procedure: labral repair
- 2 (Active Comparator): Biceps tenodesis with suture anchor
  Interventions: Procedure: biceps tenodesis
- 3 (Sham Comparator): only a diagnostic arthroscopy performed
  Interventions: Procedure: diagnostic arthroscopy

INTERVENTIONS:
Procedure: labral repair — labral repair with suture anchors
  Other Names: lupine anchor
  Arms: 1
Procedure: biceps tenodesis — biceps tenodesis with suture anchor
  Other Names: suture anchor
  Arms: 2
Procedure: diagnostic arthroscopy — diagnostic arthroscopy
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate whether there is a difference between conservative and operative treatment of Superior Labral Lesions(SLAP)of the shoulder.

DETAILED DESCRIPTION:
Treatment of superior labral lesions is controversial. Some authors advocate labral repair, some advocate biceps tenodesis,and others again questions whether these lesions should be repaired at all. There are no randomized studies comparing operative treatment and conservative treatment(i.e. physical rehabilitation), and likewise no randomized studies comparing labral repair and biceps tenodesis.

In this study;all patients who have a patient history, clinical signs of a SLAP lesion,a MRI study revealing an isolated superior labral lesion and have agreed to participate in the study, will have a diagnostic arthroscopy performed.

If a SLAP lesion is diagnosed, the patients are randomized to three different groups:1) SLAP repair with suture anchors 2) Biceps tenodesis 3) Physical therapy

ELIGIBILITY:
Inclusion Criteria:

* Clinical history and signs of superior labral lesion
* MRI study revealing an isolated superior labral lesion

Exclusion Criteria:earlier shoulder procedures,

* Other accompanying shoulderpathologies(such as cufflesions, instability, ac-joint pain, arthritis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
WOSI score Constant score EQ-5D Rowe score Patient Satisfaction | 6 and 24 months

SECONDARY OUTCOMES:
Sick leave Time back to sports at preoperative level | 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: cecilie p schrøder, MD, Principal Investigator — Lovisenberg Diakonale Hospital; Jens i Brox, MD, PhD, Study Chair — University of Oslo, Rikshospitalet
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Brox JI, Skare O, Mowinckel P, Brox JS, Reikeras O, Schroder CP. Sick leave and return to work after surgery for type II SLAP lesions of the shoulder: a secondary analysis of a randomised sham-controlled study. BMJ Open. 2020 Apr 1;10(4):e035259. doi: 10.1136/bmjopen-2019-035259. PMID 32241790
- [Derived] Schroder CP, Skare O, Reikeras O, Mowinckel P, Brox JI. Sham surgery versus labral repair or biceps tenodesis for type II SLAP lesions of the shoulder: a three-armed randomised clinical trial. Br J Sports Med. 2017 Dec;51(24):1759-1766. doi: 10.1136/bjsports-2016-097098. Epub 2017 May 11. PMID 28495804
- [Derived] Skare O, Schroder CP, Reikeras O, Mowinckel P, Brox JI. Efficacy of labral repair, biceps tenodesis, and diagnostic arthroscopy for SLAP lesions of the shoulder: a randomised controlled trial. BMC Musculoskelet Disord. 2010 Oct 7;11:228. doi: 10.1186/1471-2474-11-228. PMID 20929552